CLINICAL TRIAL: NCT02514070
Title: Comparison of EPA and DHA-Rich Fish Oils on Lipoprotein Metabolism In Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 150173; 15-H-0173
Record Dates: First submitted 2015-07-31; First posted 2015-08-03 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2019-07-24

CONDITIONS: Lipoprotein Metabolism; PCSK9; Proteomics
Keywords: LDL-C; Omega-3 Fatty Acid; PCSK9; HDL-C
MeSH Terms: interventions — Eicosapentaenoic Acid; Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- EPA-rich fish oil arm then DHA-rich fish oil arm (Experimental): Subjects randomized to the EPA-rich fish oil arm will take the equivalent to 3g of EPA /day (12 gel capsules/day) for 6 more or less 1 weeks and cross-over to the DHA-rich capsule arm
  Interventions: Drug: EPA-rich fish oil
- DHA-rich fish oil arm then EPA-rich fish oil arm (Experimental): Subjects randomized to the DHA-rich fish oil arm will take the equivalent to 3g of DHA /day (12 gel capsules/day) for 6 more or less 1 weeks and cross-over to the EPA-rich capsule arm
  Interventions: Drug: DHA-rich fish oil

INTERVENTIONS:
Drug: EPA-rich fish oil — 4 gel capsules, 3 times/day for 6 weeks
  Other Names: Eicosapentaenoic acid (EPA) Fish Oil
  Arms: EPA-rich fish oil arm then DHA-rich fish oil arm
Drug: DHA-rich fish oil — 4 gel capsules, 3 times/day for 6 weeks
  Other Names: Docosahexaenoic acid (DHA) Fish Oil
  Arms: DHA-rich fish oil arm then EPA-rich fish oil arm

SUMMARY:
Background:

- Metabolism is what the body does to turn food into energy. Omega-3 fatty acids are substances found in foods such as cold-water fish and shellfish that are essential for good health. Researchers want to see the effect of two fatty acids eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) on metabolism. They may be beneficial to cardiovascular health.

Objective:

- To understand the effects of EPA and DHA on metabolism.

Eligibility:

- Healthy people ages 18 years or above with plasma triglyceride (a type of fat in the blood) levels of 100 mg/dL or higher

Design:

* The study will last 20 to 24 weeks.
* Participants will have 4 visits to the NIH Clinical Center. These will include:
* Medical history
* Physical Fasting blood and urine tests
* CAVI tests: blood pressure is taken in the arms and legs, and the heart is monitored.
* Participants will take an EPA/DHA dietary supplement. They will take 4 gel capsules, 3 times a day, for 6 or 7 weeks. Then they will not take the capsules for 8 to 10 weeks (a wash-out period). They will then take the capsules again for 6 or 7 weeks.
* Participants will keep a food journal.

DETAILED DESCRIPTION:
This is a novel randomized crossover, double-blinded pilot study that aims to investigate the effects of different omega-3 fatty acids, namely EPA and DHA, on lipoprotein metabolism. Subjects will be unblinded for performance of measurements after they complete the study. Subjects will receive EPA or DHA supplements for approximately 6 weeks with a wash out period of 8 weeks between the two arms of the study. The study consists of 4 outpatient visits when laboratory or research samples and CAVI tests will be performed. A 7-day food diary, pill count, and red cell membrane n-3 levels will be monitored to assess compliance.

Serum cholesterol is transported by lipoproteins, such as VLDL, LDL and HDL, which vary in their relationship to cardiovascular risk. LDL is proatherogenic, whereas HDL is cardio-protective. Fish oil supplementation, such as EPA and DHA, has been shown to reduce triglycerides. EPA supplementation has also been shown to lower LDL-C, whereas DHA can raise both LDL-C and HDL-C. These differential effects on lipoproteins may alter the cardiovascular protection afforded by fish oil supplementation. This study will test the hypothesis that EPA and DHA may differ in their LDL-C lowering ability because of differences in how they modulate plasma PCSK9 levels, which is a major determinant of LDL-C levels. In addition, we will assess other parameters related to lipoprotein composition and function that may impact the cardioprotective effect of EPA and DHA. Other reported beneficial effects of omega-3 fatty acid supplementation, such as decreased platelet coagulability, markers of inflammation and changes in guy microbiota, will also be monitored.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male and female participants 18 years of age or above.
* Subject must be healthy, with no known history of cardiovascular disease.
* Subject understands protocol and provides written, informed consent in addition to a willingness to comply with specified follow-up evaluations.

EXCLUSION CRITERIA:

* Pregnancy, planned pregnancy (within the study period) or women currently breastfeeding.
* Subjects with weight changes greater than 20% over the past 3 months.
* Subjects planning a significant change in diet or exercise levels.
* Subjects already consuming more than 1.5 g per day of Eicosapentaenoic Acid (EPA) or Docosahexaenoic Acid (DHA) in any form.
* Subjects taking supplements or medications that affect lipoproteins for at least the past six weeks including fish oil supplements, bile-acid sequestrants, plant sterol supplements, fibrates, statins or Niacin.
* Subjects diagnosed with cancer or IBD, or that have taken diarrhea inhibitors, laxatives or prebiotics in the week before stool sampling (optional), or antibiotics within 3 months before sampling.
* Subjects taking daily aspirin or other anti-platelet or anti-coagulants agents (Plavix).
* History of prostate Cancer
* Subjects with known bleeding disorders (for example, Hemophilia)
* Known sensitivity or allergy to fish, shellfish or omega-3 fatty acids supplements
* Subjects with chronic diarrhea, gastric bypass or lap-band procedures, ostomies, bowel motility problems, or other conditions that could affect intestinal fat absorption
* Subjects with any acute and life-threatening condition, such as prior sudden cardiac arrest, acute myocardial infarction (last three months), stroke, embolism
* Liver enzymes (aspartate aminotransferase (AST) or alanine transaminase (ALT)) levels above 3x upper limit of normal
* Subjects initiating new medications or patients on multiple medications may also be excluded according to investigator discretion
* Subjects previously diagnosed with cardiac dysrhythmia
* Subjects with clinically diagnosed hepatic disease (including but not limited to auto immune disease, hepatitis and cirrhosis)
* Anticipated surgery during the study period
* Blood donation in the last 2 weeks or planned blood donation during the study
* Subjects requiring regular transfusions for any reason
* Subjects may also be excluded for any reason that may compromise their safety or the accuracy of research data.
* Subjects being treated with tamoxifen, estrogens, or progestins that have not been stable for >4 weeks.
* Subjects that thyroid stimulating hormone (TSH) levels are greater than 1.5 x Upper Limit of Normal (ULN) or clinical evidence of hypothyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2019-07-23 (Actual); Study Completion 2019-07-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo J Amar, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2015-H-0173.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 44 participants enrolled on protocol. 5 of these 44 participants were considered screen failures. 39 participants started the protocol.
Groups:
- Arm 1: EPA-rich Fish Oil Then DHA-rich Fish Oil: Eicosapentaenoic acid (EPA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks, followed by an 8-week washout period. Then docosahexaenoic acid (DHA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
- Arm 2: DHA-rich Fish Oil Then EPA-rich Fish Oil: Docosahexaenoic acid (DHA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks, followed by an 8-week washout period. Then Eicosapentaenoic acid (EPA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
Period: Weeks 0 to Week 6
Arm/Group | Arm 1: EPA-rich Fish Oil Then DHA-rich Fish Oil | Arm 2: DHA-rich Fish Oil Then EPA-rich Fish Oil
Started | 19 | 20
Completed | 17 | 16
Not Completed | 2 | 4
Period: Week 6 to Week 14 - Washout Period
Arm/Group | Arm 1: EPA-rich Fish Oil Then DHA-rich Fish Oil | Arm 2: DHA-rich Fish Oil Then EPA-rich Fish Oil
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0
Period: Week 14 to Week 20
Arm/Group | Arm 1: EPA-rich Fish Oil Then DHA-rich Fish Oil | Arm 2: DHA-rich Fish Oil Then EPA-rich Fish Oil
Started | 17 | 16
Completed | 16 | 14
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: EPA-rich Fish Oil, Then DHA-rich Fish Oil: Eicosapentaenoic acid (EPA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks, followed by an 8-week washout period. Then docosahexaenoic acid (DHA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
- Arm 2: DHA-rich Fish Oil, Then EPA-rich Fish Oil: Docosahexaenoic acid (DHA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks, followed by an 8-week washout period. Then Eicosapentaenoic acid (EPA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
- Total: Total of all reporting groups
Arm/Group | Arm 1: EPA-rich Fish Oil, Then DHA-rich Fish Oil | Arm 2: DHA-rich Fish Oil, Then EPA-rich Fish Oil | Total
Number analyzed (Participants) | 19 | 20 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 31 (10.7) | 34 (11.2) | 32 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 9 | 16
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 9 | 7 | 16
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Plasma PCSK9 Levels at Baseline and End of 6 Week Intervention
Description: Measure plasma proprotein convertase subtilisin/kexin type 9 (PCSK9) level, at baseline, after 6 weeks of Eicosapentaenoic acid (EPA) or Docosahexaenoic acid (DHA) fish oil supplementation.
Time Frame: baseline to 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Baseline: All study participants.
- EPA-rich Fish Oil: Eicosapentaenoic acid (EPA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
- DHA-rich Fish Oil Arm: Docosahexaenoic acid (DHA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
Arm/Group | Baseline | EPA-rich Fish Oil | DHA-rich Fish Oil Arm
Number analyzed (Participants) | 30 | 30 | 30
ng/mL | 13.30 (3.62) | 14.11 (4.36) | 12.44 (3.48)

2. Secondary Outcome: Plasma Levels in Triglyceride, Cholesterol, and Lipoprotein From Baseline to 6 Weeks
Description: Measure plasma levels at baseline to 6 weeks of intervention for the following: triglycerides (TG), low-density lipoprotein cholesterol (LDL-C), lipoprotein particle composition and size, and high-density lipoprotein (HDL) cholesterol efflux capacity.
Time Frame: Baseline to 6 weeks of intervention
Measure: Mean (Standard Deviation); unit: mg/dL
Groups:
- DHA-rich Fish Oil: Docosahexaenoic acid (DHA)-rich fish oil 4 capsules 3 times per day after meal for a total of 3g per day for 6 weeks.
Arm/Group | Baseline | EPA-rich Fish Oil | DHA-rich Fish Oil
Number analyzed (Participants) | 30 | 30 | 30
mg/dL
  Triglyceride (TG) | 95.3 (66.6) | 81.7 (64.2) | 82.1 (57.9)
  Total Cholesterol (TC) | 190.9 (52.7) | 191.1 (49.5) | 193.5 (54.4)
  LDL-C | 110.1 (49.6) | 111.4 (49.8) | 113.8 (52.5)
  Direct LDL-C | 115.7 (48.6) | 114.8 (51.3) | 120.6 (49.6)
  Small Dense LDL | 36.1 (19.9) | 37.3 (22.9) | 39.1 (23.6)
  LDL-TG | 13.1 (4) | 12.9 (4.3) | 12.8 (4)
  HDL-C | 62 (18.9) | 63.4 (20.2) | 63.4 (20.4)
  Direct HDL-C | 62.4 (16.8) | 60 (14.8) | 63.9 (17.7)
  ApoE-HDL | 5.6 (1.8) | 5.4 (1.6) | 5.9 (1.9)

ADVERSE EVENTS:
Time Frame: 20 weeks
Groups:
- Washout Period: 8 week washout period to occur between week 6 and week 14. No study supplement taken by subject at this time.
Arm/Group | EPA-rich Fish Oil | DHA-rich Fish Oil | Washout Period
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/37 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/37 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/37 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02514070/Prot_SAP_000.pdf